CLINICAL TRIAL: NCT02883283
Title: Epidural Loading Prior to Catheter Insertion: An Alternative to the Combined Spinal-epidural Technique?
Brief Title: Epidural Loading Prior to Catheter Insertion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was decided that this study was not feasible at our institution.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Goran Ristev, Assistant Clinical Professor of Anesthesiology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012H0314
Record Dates: First submitted 2016-05-09; First posted 2016-08-30 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Administration Methods of Labor Analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Catheter Administration (Active Comparator): Participants will receive the 10 mL epidural loading dose in 5 mL increments via the epidural catheter following catheter placement. (Current standard practice) Epidural loading dose via epidural catheter.
  Interventions: Procedure: Epidural loading dose; Device: Epidural catheter
- Epidural Needle Administration (Experimental): Participants will receive the 10 mL epidural loading dose in 5 mL increments via the epidural needle prior to catheter placement. Epidural loading dose via epidural needle.
  Interventions: Procedure: Epidural loading dose; Device: Epidural needle

INTERVENTIONS:
Procedure: Epidural loading dose — Labor epidural analgesia loading dose
Device: Epidural catheter — Epidural loading dose via epidural catheter
  Arms: Epidural Catheter Administration
Device: Epidural needle — Epidural loading dose via epidural needle
  Arms: Epidural Needle Administration

SUMMARY:
This study explores the potential for a more rapid onset of pain relief when drug administration is performed through the epidural needle, a technique of epidural loading that provides a rapid and reliable level of labor analgesia without the disadvantages of a combined spinal-epidural, and could add a valuable new tool to anesthesiologists.

DETAILED DESCRIPTION:
This study explores the potential for a more rapid onset of pain relief when drug administration is performed through the epidural needle, a technique of epidural loading that provides a rapid and reliable level of labor analgesia without the disadvantages of a combined spinal-epidural, and could add a valuable new tool to anesthesiologists. Investigators propose to conduct a single blinded, randomized controlled trial to determine if a difference exists in the speed of onset and spread of labor analgesia between patients receiving an epidural loading dose through the epidural needle or catheter.

Group 1 (Epidural Catheter Administration) participants will receive the 10 mL epidural loading dose in 5 mL increments via the epidural catheter following catheter placement (current standard practice).

Group 2 (Epidural Needle Administration ) participants will receive the 10 mL epidural loading dose in 5 mL increments via the epidural needle prior to catheter placement (experimental group).

Various parameters will be measured in the time after drug administration to evaluate blood pressure, heart rate, and fetal heart rate. Following delivery, the total anesthetic dose, total number of doses demanded, total number and dosage of rescue doses, and overall patient satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. subjects who have volunteered and consented to participation in the study upon admission to labor and delivery
2. parturients in active labor requesting epidural analgesia
3. uncomplicated pregnancy with a reassuring fetal heart tracing
4. age≥18 years

Exclusion Criteria:

1. contraindication to epidural anesthesia
2. inability to read, comprehend, and sign the informed consent form
3. fetal intrauterine growth retardation (IUGR)
4. non-reassuring fetal heart tracing
5. cervical dilation greater than 7cm
6. intra-uterine fetal demise
7. any spinal pathology or neurologic disease
8. history of chronic pain
9. incarcerated patients
10. any patient enrolled in the study in whom there is evidence of dural puncture during epidural technique (>3 attempts, presence of CSF).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01-23 (Actual)

PRIMARY OUTCOMES:
Mean VAS pain score | 20 minutes
  Mean VAS pain score will be determined 20 minutes following epidural loading, including assessments at 5, 10, 15, and 20 minutes.

SECONDARY OUTCOMES:
Analgesic level | 10, 15, and 20 minutes
  Analgesic level assessed by pinprick at 10, 15 and 20 minutes following loading
Maternal Blood Pressure | Baseline and 20 minutes
  Change in maternal blood pressure loading
Fetal Heart Rate | Baseline and 20 minutes
  Change in fetal heart rate over 20 minutes following loading
Rescue Bolus Count | During Labor
  Number of rescue bolus doses will be counted
Analgesia Satisfaction | During labor
  Overall patient satisfaction with analgesia following delivery via questionnaire
Intravascular catheter placement | During labor
  Incidence of intravascular catheter placement
Total anesthetic dose required | During Labor
  The total anesthetic dose during labor will be calculated
Maternal Heart Rate | Baseline and 20 minutes
  Change in maternal heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ristev, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No